CLINICAL TRIAL: NCT01790737
Title: A Prospective Phase II Study to Assess Immunophenotypic Remission After 3-drug Induction Followed by Randomized Stem Cell Mobilization, Autologous Stem Cell Transplantation (ASCT) and Lenalidomide Maintenance in Newly Diagnosed Multiple Myeloma
Brief Title: First Line Treatment Trial in Multiple Myeloma, Finnish Myeloma Group- Multiple Myeloma 02
Acronym: FMG-MM02
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Collaborators: Helsinki University Central Hospital (Other); Tampere University Hospital (Other); Turku University Hospital (Other Government); Oulu University Hospital (Other); Mikkeli Central Hospital (Other); Kymenlaakso Central Hospital Kotka Finland (Other); Jyväskylä Central Hospital (Other); Kanta-Häme Central Hospital (Other Government); Satakunta Central Hospital (Other); Kainuu Central Hospital, Kajaani (Other); Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KUH5101424; 2012-001051-39 (EudraCT Number)
Record Dates: First submitted 2013-02-04; First posted 2013-02-13 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Multiple Myeloma
Keywords: myeloma, stem cell mobilization, autologous stem cell transplantation; induction treatment, maintenance treatment
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Cyclophosphamide; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Cyclophosphamide plus filgrastim
  Interventions: Drug: Cyclophosphamide
- B (Active Comparator): Filgrastim
  Interventions: Drug: Filgrastim

INTERVENTIONS:
Drug: Cyclophosphamide
  Arms: A
Drug: Filgrastim
  Arms: B

SUMMARY:
The purpose of this study is to determinate the efficacy and safety of the 3-drug induction treatment (RVD; lenalidomide plus bortezomib plus dexamethasone)followed by randomized autologous stem cell mobilization, autologous stem cell transplantation and lenalidomide maintenance. Primary endpoint is the immunophenotypic remission rate.During the randomized mobilization phase two active comparator arms Cyclophosphamide (CY)2g/m2 + Granulocyte-colony stimulating factor(G-CSF) vrs G-CSF will be compared regarding efficacy, costs and safety.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* symptomatic, previously untreated International Stating System (ISS) 1-3 myeloma
* measurable disease
* WHO perf status 0-3
* eligible for ASCT

Exclusion Criteria:

* previously treated
* peripheral neuropathy gr >/= 2
* significant hepatic dysfunction
* severe cardiac dysfunction
* severe renal failure if not in dialysis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-01; Primary Completion 2018-10-10 (Actual); Study Completion 2019-02-26 (Actual)

PRIMARY OUTCOMES:
Immunophenotypic response | Change from the start of induction treatment at 3 months, change from the start of induction at 6 months, at 9 months, at 12 months, at 16 months, at 20 months, at 24 moths
  Response will be measured by International Myeloma Working Group (IMWG) guidelines, and if the response is stringent CR and immunophenotypic remission, those patients will be followed also by allele-spesific oligonucleotide-polymerase chain reaction assay (ASO-PCR) to find out molecular remission rate.

SECONDARY OUTCOMES:
Progression free survival | From date of inclusion until the date of first documented progression or date of death from any cause whatever come first assessed up to last patient 2 years on maintenance

OTHER OUTCOMES:
Proportion of pts collected with >/= 3 x 10e6/kg CD34+ with </= 2 apheresis after mobilization with CY 2g/m2 + filgrastim (group A) or filgrastim alone (group B) | Assessed up to 2 weeks from the start of mobilization

CONTACTS AND LOCATIONS:
Overall Officials: Raija Silvennoinen, MD, Principal Investigator — Kuopio University Hospital, Kuopio, FI
Locations (12):
- Finland (12):
  - Kuopio University Hospital, Kuopio, Northern Savonia
  - Tampere University Hospital, Tampere, Pirkanmaa
  - Kanta-Häme Central Hospital, Hämeenlinna
  - Helsinki University Hospital, Helsinki
  - Jyväskylä Central Finland Central Hospital, Jyväskylä
  - Kainuu Kajaani Central Hospital, Kajaani
  - Länsi-Pohja Central Hospital, Kemi
  - Kymenlaakso Central Hospital, Kotka
  - Mikkeli Southern-Savo Central Hospital, Mikkeli
  - Oulu University Hospital, Oulu
  - Satakunta Central Hospital, Pori
  - Turku University Central Hospital, Turku